CLINICAL TRIAL: NCT05066815
Title: Evaluation of Crestal Bone Loss Around Short Dental Implants As Affected By Two Suprastructure Materials
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Dina Nabil Ezz Eldin, : Assistant Lecturer of Fixed Prosthodontics, Faculty of Dentistry (Aswan University), Cairo University
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: 211020
Record Dates: First submitted 2021-08-11; First posted 2021-10-04 (Actual); Last update posted 2022-06-10 (Actual); Status verified 2022-06

CONDITIONS: Bone Loss
MeSH Terms: conditions — Bone Diseases, Metabolic | interventions — VITA Enamic

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hybrid superstructure (Experimental): screw retained hybrid ceramic crowns
  Interventions: Other: Vita Enamic (Hybrid dental ceramic)
- Ceramic superstructure (Active Comparator): screw retained lithium disilicate based ceramic crowns
  Interventions: Other: Vita Enamic (Hybrid dental ceramic)

INTERVENTIONS:
Other: Vita Enamic (Hybrid dental ceramic) — Vita Enamic (Hybrid dental ceramic) is provided as blocks to be milled using Computer aided design/Computer aided manufacturer (CAD/CAM) technology.
  Other Names: Polymer Infiltrated Ceramic Network (PICN)

SUMMARY:
The aim of the study is to evaluate the crestal bone loss developed around short dental implants after using screw retained Hybrid ceramic crowns when compare to screw retained Lithium Di silicate based ceramic crowns.

DETAILED DESCRIPTION:
This study will be conducted on patients requiring single implant replacement in the posterior regions of the mandible, admitted to the Outpatient Clinic of Fixed Prosthodontics Department, Faculty of Oral and Dental medicine, Cairo University.

Examination and diagnosis:

1. Selection and examination of the patients according to inclusion and exclusion criteria.
2. Preoperative Cone Beam Computed Tomography (CBCT) to all patients.
3. Primary impression will be taken to produce study cast.
4. Taking a professional photo for the examined posterior area.
5. Patients will be divided into two group:

G1: Short implants will be restored by screw retained Hybrid ceramic crowns G2: Short implants will be restored by screw retained Lithium Di silicate based ceramic crowns

Surgical procedures:

* Implants will be placed following standardized protocol.
* After 4 months the patients re-attended for placement of healing abutments for about (10-14) days and prosthesis fabrication.

Data collection and post operative radio-logical assessment:

-Taking standardized digital peri-apical radio-graph by paralleling technique and film holding device for follow up at 12 months after crowns loading to evaluate crestal bone loss.

ELIGIBILITY:
Inclusion Criteria:

1. Patients within age group of ≥ 18.
2. There should be absence of any systemic diseases.
3. Patients have missing simple posterior tooth
4. Adequate interarch space.
5. Inadequate residual bone height to place standard length implant.
6. Patients with good oral hygiene.

Exclusion Criteria:

1. A history that would complicate the outcome of the study, such as alcohol or drug dependency, smoking, poor health, or any other medical, physical or psychological reason that might affect the surgical procedure or the subsequent prosthodontics treatment and required follow-up.
2. Heavy smokers.
3. Poorly controlled diabetes mellitus.
4. Patients on radiotherapy.
5. Patients with temporomandibular disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-10-25 (Estimated); Primary Completion 2022-12-25 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Crestal Bone Loss Crestal bone loss will be measured using standardized digital periapical radiograph by paralleling technique and film holding device -measuring unit:Milimeters | one year
  preventive

SECONDARY OUTCOMES:
screw loosening of crowns screw loosening will be observed by clinical investigation -measuring unit:Binary (Yes/No) | one year
  preventive